CLINICAL TRIAL: NCT04057937
Title: A Phase 2, Multi-Center, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Evaluate the Efficacy and Safety of Apremilast (CC-10004) in the Treatment of Palmoplantar Pustulosis in Japan
Brief Title: A Study to Evaluate the Efficacy and Safety of Apremilast (CC-10004) in Japanese Subjects With Palmoplantar Pustulosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CC-10004-PPP-001; U1111-1236-1239 (Other: WHO)
Record Dates: First submitted 2019-08-13; First posted 2019-08-15 (Actual); Results first posted 2022-01-06 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Palmoplantaris Pustulosis
Keywords: Palmoplantar Pustulosis; CC-10004; Apremilast; Only Japanese; Efficacy; Safety; Phase 2
MeSH Terms: conditions — Psoriasis | interventions — apremilast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Placebo then Apremilast 30mg BID (Experimental): Participants received matched placebo as oral tablets twice daily (BID) for up to 16 weeks (Week 0 to Week 16). Participants who completed the placebo-controlled phase entered the active-treatment phase and received apremilast 30 mg as oral tablets BID for up to an additional 16 weeks (Week 16 to Week 32).
  Interventions: Drug: Apremilast; Drug: Placebo
- Apremilast 30 mg BID then Apremilast 30 mg BID (Experimental): Participants received apremilast 30 mg as oral tablets BID for up to 16 weeks (Week 0 to Week 16). Participants who completed the placebo-controlled phase entered the active-treatment phase and received apremilast 30 mg as oral tablets BID for up to an additional 16 weeks (Week 16 to Week 32).
  Interventions: Drug: Apremilast

INTERVENTIONS:
Drug: Apremilast — Apremilast
  Other Names: CC-10004
Drug: Placebo — Placebo
  Arms: Placebo then Apremilast 30mg BID

SUMMARY:
This study will evaluate whether apremilast is better than placebo (inactive substance in the same form as the drug) for the treatment in Japanese subjects with PPP. This study also will evaluate the safety and tolerability of apremilast in Japanese subjects with PPP.CC-10004-PPP-001 is a multicenter, randomized, double-blind, placebo-controlled, parallel group, Phase 2 study of apremilast in Japanese subjects with PPP and inadequate response to treatment with topical steroid and/or topical vitamin D3 derivative preparations.

The placebo-controlled period will be 16 weeks and patients will receive apremilast or placebo. After the 16-week placebo-controlled period, all subjects will receive apremilast for 16 weeks. All subjects will have their final study visit 4 weeks after stopping apremilast treatment.

ELIGIBILITY:
Inclusion Criteria:

Subjects must satisfy the following criteria to be enrolled in the study:

1. Subject has a diagnosis of Palmoplantar Pustulosis with or without pustulotic arthro-osteitis (PAO) for at least 24 weeks before screening.
2. Subject has a total score of PPPASI: ≥ 12 at screening and baseline.
3. Subject has moderate or severe pustules/vesicles on palms or soles (PPPASI severity score: ≥ 2) at screening and baseline.
4. Subject has inadequate response to treatment with topical steroid and/or topical vitamin D3 derivative preparations prior to or at screening.

Exclusion Criteria:

The presence of any of the following will exclude a subject from enrollment:

1. Subject has a diagnosis of plaque-type psoriasis.
2. Subject has the presence of pustular psoriasis in any part of the body other than the palms and soles.
3. Subject has obvious improvement during screening (≥ 5 PPPASI total score improvement during the screening).
4. Subject has received any procedures for focal infection (e.g, tonsillectomy and dental therapy) within 24 weeks of baseline.
5. Subject has periodontitis obviously requiring treatment at screening.
6. Subject has chronic or recurrent tonsillitis or sinusitis requiring any continuous treatment for a month or more at screening.
7. Subject has evidence of skin conditions of hands and feet that would interfere with evaluations of the effect of study medication.
8. Subject is pregnant or breastfeeding.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2019-10-16 (Actual); Primary Completion 2021-01-18 (Actual); Study Completion 2021-06-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (22):
- Japan (22):
  - Research Site, Ichinomiya, Aichi-ken
  - Research Site, Nagoya, Aichi-ken
  - Research Site, Fukuoka, Fukuoka
  - Research Site, Sapporo, Hokkaido
  - Research Site, Hitachi, Ibaraki
  - Research Site, Sagamihara-shi, Kanagawa
  - Research Site, Yokohoma-shi, Kanagawa
  - Research Site, Yokosuka, Kanagawa
  - Research Site, Izumo, Shimane
  - Research Site, Chiyoda-ku, Tokyo
  - Research Site, Itabashi-ku, Tokyo
  - Research Site, Itabashi-ku
  - Research Site, Kisarazu
  - Research Site, Kofu
  - Research Site, Minokamo
  - Research Site, Nankoku-shi
  - Research Site, Osaka
  - Research Site, Sendai
  - Research Site, Shinjuku-ku
  - Research Site, Shinjyuku-ku
  - Research Site, Tōon
  - Research Site, Tsu

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- [Background] Terui T, Okubo Y, Kobayashi S, Sano S, Morita A, Imafuku S, Tada Y, Abe M, Yaguchi M, Uehara N, Handa T, Tanaka M, Zhang W, Paris M, Murakami M. Efficacy and Safety of Apremilast for the Treatment of Japanese Patients with Palmoplantar Pustulosis: Results from a Phase 2, Randomized, Placebo-Controlled Study. Am J Clin Dermatol. 2023 Sep;24(5):837-847. doi: 10.1007/s40257-023-00788-2. Epub 2023 May 26. PMID 37233897
- [Background] Okubo Y, Terui T, Kobayashi S, Sano S, Morita A, Imafuku S, Tada Y, Abe M, Yaguchi M, Kimura T, Shimauchi J, Zhang W, Amouzadeh H, Murakami M. Exploratory Efficacy Evaluation of Apremilast for the Treatment of Japanese Patients with Palmoplantar Pustulosis: 32-Week Results from a Phase 2, Randomized, Placebo-Controlled Study. Dermatol Ther (Heidelb). 2024 Jul;14(7):1863-1873. doi: 10.1007/s13555-024-01195-z. Epub 2024 Jun 19. PMID 38896381
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Japanese participants with palmoplantar pustulosis (PPP) were enrolled at 22 research centers in Japan from October 2019 to June 2021.
Pre-assignment Details: Participants were randomized in a 1:1 ratio to receive either apremilast or matched placebo from Week 0 to Week 16 (placebo-controlled phase) of the study. Eligible participants then entered an active-treatment phase and received apremilast from after Week 16 to Week 32.
Groups:
- Placebo Then Apremilast 30mg BID: Participants received matched placebo as oral tablets twice daily (BID) for up to 16 weeks (Week 0 to Week 16). Participants who completed the placebo-controlled phase entered the active-treatment phase and received apremilast 30 mg as oral tablets BID for up to an additional 16 weeks (after Week 16 to Week 32).
- Apremilast 30 mg BID Then Apremilast 30 mg BID: Participants received apremilast 30 mg as oral tablets BID for up to 16 weeks (Week 0 to Week 16). Participants who completed the placebo-controlled phase entered the active-treatment phase and received apremilast 30 mg as oral tablets BID for up to an additional 16 weeks (after Week 16 to Week 32).
Period: Placebo-controlled Phase
Arm/Group | Placebo Then Apremilast 30mg BID | Apremilast 30 mg BID Then Apremilast 30 mg BID
Started | 44 | 46
Completed | 41 | 46
Not Completed | 3 | 0
Not completed — Adverse Event | 3 | 0
Period: Active-treatment Phase
Arm/Group | Placebo Then Apremilast 30mg BID | Apremilast 30 mg BID Then Apremilast 30 mg BID
Started | 41 | 46
Completed | 40 | 44
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Pregnancy | 0 | 1
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Then Apremilast 30mg BID | Apremilast 30 mg BID Then Apremilast 30 mg BID | Total
Number analyzed (Participants) | 44 | 46 | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.7 (11.68) | 54.9 (11.30) | 54.8 (11.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 36 | 69
  Male | 11 | 10 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 44 | 46 | 90
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 44 | 46 | 90
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Palmo-plantar Pustulosis Area and Severity Index (PPPASI) Score [Mean (Standard Deviation); unit: Score on a scale] — PPPASI is a disease-specific efficacy assessment tool to evaluate for 3 signs of the disease (erythema, pustules/vesicle and desquamation/scale) as sub-scores on palms or soles. The PPPASI total scores are calculated by sum of the sub-scores and range from 0 to 72 with a higher score indicating more severe disease.
  Score on a scale | 24.93 (8.915) | 25.03 (8.675) | 24.98 (8.744)
Palmo-plantar Severity Index (PPSI) Total Score [Mean (Standard Deviation); unit: Score on a Scale] — PPSI is a disease-specific assessment tool for grading the severity of PPP lesions. Evaluation of skin lesion sites are assessed separately for erythema, pustules/vesicle and desquamation/scale, which are each rated on a scale of 0 to 4. The PPSI produces a total numeric score that ranges from 0 to 12. A higher score indicates more severe disease.
  Score on a Scale | 8.2 (1.49) | 8.3 (1.48) | 8.20 (1.48)
Physician's Global Assessment (PGA) Score for Palms and Soles [Count of Participants; unit: Participants] — The PGA for palms and soles is used to determine the participants' PPP lesions on palms and soles. Lesions on palms and soles are graded from 0-5 with a higher score indicating more severe disease. The number of participants with each of the PGA score categories at baseline are reported:
  0 = Clear
  1. = Almost clear/Minimal
  2. = Mild
  3. = Moderate
  4. = Severe
  5. = Very severe
  Participants
    0 = Clear | 0 | 0 | 0
    1 = Almost clear/Minimal | 0 | 0 | 0
    2 = Mild | 1 | 3 | 4
    3 = Moderate | 24 | 16 | 40
    4 = Severe | 17 | 21 | 38
    5 = Very severe | 2 | 6 | 8
Participants Visual Analogue Scale (VAS) Assessment for PPP Symptoms [Mean (Standard Deviation); unit: Score on a Scale] — Participants assessed the degree of both pruritus itching and skin discomfort/pain as symptoms on hands and feet caused by PPP on a VAS. Each score ranges from 0 to 100. The left-hand boundary (0) on the VAS represents no itch/pain and the right-hand boundary (100) represents itch/pain as severe as can be imagined by the participant. Population: VAS assessment was missed by 2 participants in the placebo arm at baseline.
  Score on a Scale
    Itching: number analyzed (Participants) | 42 | 46 | 88
    Itching | 57.0 (27.8) | 50.3 (31.58) | 53.5 (29.85)
    Discomfort/Pain: number analyzed (Participants) | 42 | 46 | 88
    Discomfort/Pain | 50.3 (29.98) | 45.4 (31.92) | 47.8 (30.93)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieve a PPPASI-50 at Week 16
Description: PPPASI-50 is defined as >= 50 percent decrease in PPPASI total score from baseline.
  PPPASI is a disease-specific efficacy assessment tool to evaluated for 3 signs of the disease (erythema, pustules/vesicle and desquamation/scale) as sub-scores on palms or soles. The PPPASI total scores are calculated by sum of the sub-scores and range from 0 to 72 with a higher score indicating more severe disease.
Time Frame: At Week 16
Population: Intent-to-treat (ITT) population which includes all randomized participants who received at least one dose of investigational product.
Measure: Number; unit: Percentage of Partcipants
Groups:
- Placebo-controlled Phase - Placebo: Participants received matched placebo as oral tablets BID for up to 16 weeks (Week 0 to Week 16).
- Placebo-controlled Phase - Apremilast 30 mg BID: Participants received apremilast 30 mg as oral tablets BID for up to 16 weeks (Week 0 to Week 16).
Arm/Group | Placebo-controlled Phase - Placebo | Placebo-controlled Phase - Apremilast 30 mg BID
Number analyzed (Participants) | 44 | 46
Percentage of Partcipants | 40.9 | 78.3
Statistical Analysis 1: Comparison: Placebo-controlled Phase - Placebo vs Placebo-controlled Phase - Apremilast 30 mg BID; Test type: Superiority; p = 0.0003, Chi-squared — Two-sided 0.10 significant level; Percentage Difference:Apremilast-Placebo = 37.4, 95% CI 2-sided [18.6 to 56.1] — Confidence Intervals calculated using the Wald method (normal approximation)

2. Secondary Outcome: Percentage of Participants Who Achieve a PPPASI-50 at All Other Visits in Placebo-controlled Phase
Description: PPPASI-50 is defined as >= 50 percent decrease in PPPASI total score from baseline.
  PPPASI is a disease-specific efficacy assessment tool to evaluated for 3 signs of the disease (erythema, pustules/vesicle and desquamation/scale) as sub-scores on palms or soles. The PPPASI total scores are calculated by sum of the sub-scores and range from 0 to 72 with a higher score indicating more severe disease. Missing values at were imputed using non-responder imputation (NRI) as the primary method, by which a participant without sufficient data for the response determination was considered a non-responder.
Time Frame: Weeks 2 to 14
Population: ITT population which includes all randomized participants who received at least one dose of investigational product.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo-controlled Phase - Placebo | Placebo-controlled Phase - Apremilast 30 mg BID
Number analyzed (Participants) | 44 | 46
Percentage of Participants
  Week 2 | 2.3 | 30.4
  Week 4 | 18.2 | 52.2
  Week 6 | 18.2 | 69.6
  Week 8 | 43.2 | 65.2
  Week 10 | 34.1 | 71.7
  Week 12 | 34.1 | 69.6
  Week 14 | 47.7 | 73.9

3. Secondary Outcome: Percentage of Participants Who Achieve a PPPASI-75 at Each Visit in Placebo-controlled Phase
Description: PPPASI-75 is defined as >=75 percent decrease in PPPASI total score from baseline.
  PPPASI is a disease-specific efficacy assessment tool to evaluated for 3 signs of the disease (erythema, pustules/vesicle and desquamation/scale) as sub-scores on palms or soles. The PPPASI total scores are calculated by sum of the sub-scores and range from 0 to 72 with a higher score indicating more severe disease. Missing values were imputed using NRI as the primary method, by which a participant without sufficient data for the response determination was considered a non-responder.
Time Frame: Weeks 2 to 16
Population: ITT population which includes all randomized participants who received at least one dose of investigational product.
Measure: Number; unit: Percentage of Partcipants
Arm/Group | Placebo-controlled Phase - Placebo | Placebo-controlled Phase - Apremilast 30 mg BID
Number analyzed (Participants) | 44 | 46
Percentage of Partcipants
  Week 2 | 2.3 | 2.2
  Week 4 | 4.5 | 10.9
  Week 6 | 9.1 | 21.7
  Week 8 | 11.4 | 19.6
  Week 10 | 11.4 | 30.4
  Week 12 | 13.6 | 30.4
  Week 14 | 13.6 | 37.0
  Week 16 | 15.9 | 43.5

4. Secondary Outcome: Area Under the Curve (AUC) of PPPASI Total Score From Baseline Through Week 16
Description: The AUC for PPPASI total score from baseline through Week 16 is the sum of the AUCs in each time interval specified by the dates of the visits and is calculated based on the linear trapezoidal method.
  PPPASI is a disease-specific efficacy assessment tool to evaluate 3 signs of the disease (erythema, pustules/vesicle and desquamation/scale) as sub-scores on palms or soles. The PPPASI total scores are calculated by sum of the sub-scores and range from 0 to 72 with a higher score indicating more severe disease.
Time Frame: Baseline to Week 16
Population: ITT population which includes all randomized participants who received at least one dose of investigational product.
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores * Day
Arm/Group | Placebo-controlled Phase - Placebo | Placebo-controlled Phase - Apremilast 30 mg BID
Number analyzed (Participants) | 44 | 46
Scores * Day | 1911.74 [1707.92 to 2115.57] | 1337.49 [1134.52 to 1540.47]

5. Secondary Outcome: Percent Change From Baseline in PPPASI Total Score by Visit in Placebo-controlled Phase .
Description: PPPASI is a disease-specific efficacy assessment tool to evaluated for 3 signs of the disease (erythema, pustules/vesicle and desquamation/scale) as sub-scores on palms or soles. The PPPASI total scores are calculated by sum of the sub-scores and range from 0 to 72 with a higher score indicating more severe disease. A positive change from baseline indicates a worsening of symptoms.
Time Frame: Baseline to Week 16
Population: ITT population which includes all randomized participants who received at least one dose of investigational product. Only participants with data available for analysis are reported.
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Placebo-controlled Phase - Placebo | Placebo-controlled Phase - Apremilast 30 mg BID
Number analyzed (Participants) | 44 | 46
Percent Change
  Week 2 | -11.09 (22.102) | -36.62 (22.816)
  Week 4: number analyzed (Participants) | 43 | 46
  Week 4 | -23.82 (28.307) | -48.96 (21.973)
  Week 6: number analyzed (Participants) | 43 | 46
  Week 6 | -30.15 (24.826) | -55.06 (23.164)
  Week 8: number analyzed (Participants) | 43 | 46
  Week 8 | -42.41 (27.115) | -57.11 (22.710)
  Week 10: number analyzed (Participants) | 42 | 46
  Week 10 | -36.52 (32.999) | -60.85 (21.792)
  Week 12: number analyzed (Participants) | 41 | 46
  Week 12 | -42.30 (26.802) | -61.22 (22.787)
  Week 14: number analyzed (Participants) | 41 | 46
  Week 14 | -45.00 (30.915) | -63.78 (23.952)
  Week 16: number analyzed (Participants) | 41 | 46
  Week 16 | -42.35 (32.671) | -64.33 (24.345)

6. Secondary Outcome: Change From Baseline in PPPASI Total Score at Week 16
Description: PPPASI is a disease-specific efficacy assessment tool to evaluated for 3 signs of the disease (erythema, pustules/vesicle and desquamation/scale) as sub-scores on palms or soles. The PPPASI total scores are calculated by sum of the sub-scores and range from 0 to 72 with a higher score indicating more severe disease. Change from baseline based on a mixed-effects model for repeated measures with a positive change indicating a worsening of symptoms.
Time Frame: Baseline and Week 16
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo-controlled Phase - Placebo | Placebo-controlled Phase - Apremilast 30 mg BID
Number analyzed (Participants) | 41 | 46
Units on a scale | -11.03 (1.260) | -16.48 (1.224)

7. Secondary Outcome: AUC for PPSI Total Score From Baseline Through Week 16
Description: The AUC for PPSI total score from baseline through Week 16 is the sum of the AUCs in each time interval specified by the dates of the visits and is calculated based on the linear trapezoidal method. PPSI is a disease-specific assessment tool for grading the severity of PPP lesions. Evaluation of skin lesion sites are assessed separately for erythema, pustules/vesicle and desquamation/scale, which are each rated on a scale of 0 to 4. The PPSI produces a total numeric score that ranges from 0 to 12. A higher score indicates more severe disease.
Time Frame: Baseline to Week 16
Population: ITT population which includes all randomized participants who received at least one dose of investigational product.
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores * Day
Arm/Group | Placebo-controlled Phase - Placebo | Placebo-controlled Phase - Apremilast 30 mg BID
Number analyzed (Participants) | 44 | 46
Scores * Day | 725.62 [668.09 to 783.15] | 564.63 [507.35 to 621.90]

8. Secondary Outcome: Percent Change From Baseline in PPSI Total Score by Visit in Placebo-controlled Phase
Description: PPSI is a disease-specific assessment tool for grading the severity of PPP lesions. Evaluation of skin lesion sites are assessed separately for erythema, pustules/vesicle and desquamation/scale, which are each rated on a scale of 0 to 4. The PPSI produces a total numeric score that ranges from 0 to 12. A higher score indicates more severe disease. A positive change from baseline indicates a worsening of symptoms.
Time Frame: Baseline to Week 16
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Placebo-controlled Phase - Placebo | Placebo-controlled Phase - Apremilast 30 mg BID
Number analyzed (Participants) | 44 | 46
Percent Change
  Week 2 | -6.25 (19.409) | -24.70 (19.780)
  Week 4: number analyzed (Participants) | 43 | 46
  Week 4 | -13.84 (25.629) | -34.58 (23.190)
  Week 6: number analyzed (Participants) | 43 | 46
  Week 6 | -20.02 (20.639) | -40.50 (23.035)
  Week 8: number analyzed (Participants) | 43 | 46
  Week 8 | -30.12 (29.340) | -40.76 (23.019)
  Week 10: number analyzed (Participants) | 42 | 46
  Week 10 | -27.42 (29.635) | -44.22 (24.890)
  Week 12: number analyzed (Participants) | 41 | 46
  Week 12 | -31.18 (27.817) | -46.47 (25.202)
  Week 14: number analyzed (Participants) | 41 | 46
  Week 14 | -34.98 (28.205) | -50.16 (25.488)
  Week 16: number analyzed (Participants) | 41 | 46
  Week 16 | -30.90 (25.414) | -48.96 (21.821)

9. Secondary Outcome: Change From Baseline in PPSI Total Score at Week 16
Description: PPSI is a disease-specific assessment tool for grading the severity of PPP lesions. Evaluation of skin lesion sites are assessed separately for erythema, pustules/vesicle and desquamation/scale, which are each rated on a scale of 0 to 4. The PPSI produces a total numeric score that ranges from 0 to 12. A higher score indicates more severe disease. Change from baseline based on a mixed-effects model for repeated measures with a positive change indicating a worsening of symptoms.
Time Frame: Baseline and Week 16
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo-controlled Phase - Placebo | Placebo-controlled Phase - Apremilast 30 mg BID
Number analyzed (Participants) | 41 | 46
Units on a scale | -2.56 (0.303) | -4.19 (0.293)

10. Secondary Outcome: Percentage of Participants Achieving a PGA Score of Clear (0) or Minimal (1) by Visit in Placebo-controlled Phase
Description: The PGA for palms and soles was used to determine the participants PPP lesions on palms and soles. Lesions on palms and soles were graded based on the following scales:
  0 = Clear
  1. = Almost clear/Minimal
  2. = Mild
  3. = Moderate
  4. = Severe
  5. = Very severe.
  The percentage of of participants with a post baseline score of 0 or 1 (responders) are reported. Missing values at were imputed using NRI as the primary method, by which a participant without sufficient data for the response determination was considered a non-responder.
Time Frame: Weeks 2 to 16
Population: ITT population which includes all randomized participants who received at least one dose of investigational product. Only participants with a PGA greater than 1 at baseline are included in this analysis.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo-controlled Phase - Placebo | Placebo-controlled Phase - Apremilast 30 mg BID
Number analyzed (Participants) | 44 | 46
Percentage of Participants
  Week 2 | 0.0 | 2.2
  Week 4 | 2.3 | 4.3
  Week 6 | 2.3 | 4.3
  Week 8 | 9.1 | 8.7
  Week 10 | 9.1 | 13.0
  Week 12 | 9.1 | 15.2
  Week 14 | 9.1 | 17.4
  Week 16 | 4.5 | 19.6

11. Secondary Outcome: Percentage of Participants Achieving a PGA Score of 0 or 1 With At Least a 2 Grade Improvement by Visit in Placebo-controlled Phase.
Description: The PGA for palms and soles was used to determine the participants PPP lesions on palms and soles. Lesions on palms and soles were graded based on the following scales:
  0 = Clear
  1. = Almost clear/Minimal
  2. = Mild
  3. = Moderate
  4. = Severe
  5. = Very severe.
  The percentage of of participants with at least a 2 grade improvement from baseline (stringent responders) are reported. issing values at were imputed using NRI as the primary method, by which a participant without sufficient data for the response determination was considered a non-responder.
Time Frame: Weeks 2 to 16
Population: as for outcome 10
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo-controlled Phase - Placebo | Placebo-controlled Phase - Apremilast 30 mg BID
Number analyzed (Participants) | 44 | 46
Percentage of Participants
  Week 2 | 0.0 | 2.2
  Week 4 | 2.3 | 4.3
  Week 6 | 2.3 | 4.3
  Week 8 | 9.1 | 6.5
  Week 10 | 9.1 | 10.9
  Week 12 | 9.1 | 15.2
  Week 14 | 9.1 | 17.4
  Week 16 | 4.5 | 17.4

12. Secondary Outcome: Change From Baseline in Participant VAS Assessment for PPP Symptoms
Description: Participants assessed the degree of both pruritus itching and skin discomfort/pain as symptoms on hands and feet caused by PPP on a VAS. Each score ranged from 0 to 100. The left-hand boundary (0) on the VAS represents no itch/pain and the right-hand boundary (100) represents itch/pain as severe as can be imagined by participant.
Time Frame: Baseline and Weeks 2,4,6,8,12,16
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on scale
Arm/Group | Placebo-controlled Phase - Placebo | Placebo-controlled Phase - Apremilast 30 mg BID
Number analyzed (Participants) | 42 | 46
Units on scale
  Itching Week 2: number analyzed (Participants) | 41 | 43
  Itching Week 2 | -2.4 (25.07) | -25.0 (24.42)
  Itching Week 4: number analyzed (Participants) | 39 | 43
  Itching Week 4 | -7.9 (21.39) | -22.7 (26.36)
  Itching Week 6: number analyzed (Participants) | 40 | 43
  Itching Week 6 | -9.3 (29.65) | -22.4 (29.37)
  Itching Week 8: number analyzed (Participants) | 40 | 43
  Itching Week 8 | -19.0 (25.53) | -24.8 (29.38)
  Itching Week 12: number analyzed (Participants) | 38 | 43
  Itching Week 12 | -14.9 (35.82) | -28.3 (28.55)
  Itching Week 16: number analyzed (Participants) | 38 | 43
  Itching Week 16 | -10.5 (30.81) | -26.8 (28.65)
  Discomfort/Pain Week 2: number analyzed (Participants) | 42 | 43
  Discomfort/Pain Week 2 | -0.7 (32.47) | -20.2 (26.73)
  Discomfort/Pain Week 4: number analyzed (Participants) | 40 | 43
  Discomfort/Pain Week 4 | -6.9 (30.39) | -21.6 (29.21)
  Discomfort/Pain Week 6: number analyzed (Participants) | 41 | 43
  Discomfort/Pain Week 6 | -6.7 (28.80) | -22.4 (33.16)
  Discomfort/Pain Week 8: number analyzed (Participants) | 41 | 43
  Discomfort/Pain Week 8 | -15.5 (31.14) | -22.0 (29.02)
  Discomfort/Pain Week 12: number analyzed (Participants) | 39 | 43
  Discomfort/Pain Week 12 | -14.1 (32.07) | -27.6 (28.14)
  Discomfort/Pain Week 16: number analyzed (Participants) | 39 | 43
  Discomfort/Pain Week 16 | -13.5 (27.51) | -25.3 (29.51)

ADVERSE EVENTS:
Time Frame: Placebo-controlled Phase: Week 0 to Week 16. Active-treatment Phase: After Week 16 to Week 32.
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold
Groups:
- Active-treatment Phase - Apremilast 30 mg BID: All participants who completed the placebo-controlled phase entered the active-treatment phase and received apremilast 30 mg as oral tablets BID for up to an additional 16 weeks (after Week 16 to Week 32).
Arm/Group | Placebo-controlled Phase - Placebo | Placebo-controlled Phase - Apremilast 30 mg BID | Active-treatment Phase - Apremilast 30 mg BID
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/46 | 0/87
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/46 | 3/87
Other Adverse Events (participants affected / at risk) | 16/44 | 32/46 | 40/87
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo-controlled Phase - Placebo (N=44) | Placebo-controlled Phase - Apremilast 30 mg BID (N=46) | Active-treatment Phase - Apremilast 30 mg BID (N=87)
Constipation (Gastrointestinal disorders) | 0 | 0 | 1
Volvulus (Gastrointestinal disorders) | 0 | 0 | 1
COVID-19 pneumonia (Infections and infestations) | 0 | 0 | 1
Peritonitis (Infections and infestations) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo-controlled Phase - Placebo (N=44) | Placebo-controlled Phase - Apremilast 30 mg BID (N=46) | Active-treatment Phase - Apremilast 30 mg BID (N=87)
Abdominal discomfort (Gastrointestinal disorders) | 1 | 7 | 6
Diarrhoea (Gastrointestinal disorders) | 6 | 12 | 8
Faeces soft (Gastrointestinal disorders) | 2 | 5 | 3
Nausea (Gastrointestinal disorders) | 2 | 6 | 3
Folliculitis (Infections and infestations) | 4 | 1 | 3
Nasopharyngitis (Infections and infestations) | 2 | 5 | 5
Decreased appetite (Metabolism and nutrition disorders) | 0 | 3 | 1
Headache (Nervous system disorders) | 0 | 6 | 4
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 5 | 5
Eczema (Skin and subcutaneous tissue disorders) | 5 | 3 | 3
Pustulotic arthro-osteitis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 5
Palmoplantar pustulosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2020-04-20): https://cdn.clinicaltrials.gov/large-docs/37/NCT04057937/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-04): https://cdn.clinicaltrials.gov/large-docs/37/NCT04057937/SAP_001.pdf